CLINICAL TRIAL: NCT04003818
Title: Prospective, Interventional, Phase IV Study, Evaluating the Efficacy and Safety of Teicoplanin (100-200 mg, Administered Orally Twice a Day) in Patients With Clostridium Difficile Infection-associated Diarrhea and Colitis
Brief Title: Efficacy and Safety of Teicoplanin in CDAD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to COVID-19 and great challenges during patient enrolment period, current status of this study is far behind the plan. The study cannot be completed according to the plan. Sanofi decides to terminate the study upon comprehensive assessment.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16229; U1111-1230-0601 (Other: UTN)
Record Dates: First submitted 2019-06-06; First posted 2019-07-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Clostridium Difficile Infection-associated Diarrhea and Colitis
MeSH Terms: conditions — Colitis | interventions — Teicoplanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Teicoplanin (Experimental): teicoplanin, administered orally 100-200 mg, twice a day
  Interventions: Drug: TEICOPLANIN

INTERVENTIONS:
Drug: TEICOPLANIN — Pharmaceutical form:solution for oral administration Route of administration: oral

SUMMARY:
Primary Objective:

Explore the efficacy of teicoplanin (100-200 mg administered orally twice a day for 7 to 14 days) in patients with Clostridium difficile infection-associated diarrhea and colitis

Secondary Objective:

Evaluate the safety of teicoplanin in patients with Clostridium difficile infection-associated diarrhea and colitis

DETAILED DESCRIPTION:
Approximate 10 weeks

ELIGIBILITY:
Inclusion criteria :

* Signed Informed Consent.
* Male or female no less than 18 years of age.
* Inpatient with a diagnosis of mild-moderate or severe CDAD (first occurrence or first recurrence within 3 months) with: Diarrhea: a change in bowel habits with > 3 liquid or unformed bowel movements (UBM) within 24 hours prior to enrollment, AND Positive C. difficile toxin test on a stool sample produced within 72 hours prior to enrollment.

Exclusion criteria:

* More than one previous episode of CDAD in the 3-month period prior to enrollment.
* Evidence of life-threatening or fulminant CDAD.
* Likelihood of death within 72 hours from any cause.
* History of inflammatory colitides, chronic abdominal pain, or chronic diarrhea
* Antimicrobial treatment active against CDAD administered for > 24 hours except for metronidazole treatment failures (MTF).
* Known hypersensitivity or contraindication to teicoplanin.
* Pregnant or nursing females.
* Unable or unwilling to comply with all protocol requirements.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate | 2 days after 7-14 days treatment
  Clinical cure is defined as: Resolution of diarrhea (ROD) (≤ 3 unformed bowel movement (UBM) per day for at least 2 consecutive days) on study treatment and maintained for 2 days after End of treatment (EOT), AND No additional antimicrobial treatment active against Clostridium difficile-associated diarrhea (CDAD) or fecal microbiota transplant (FMT) between first dose of study drug and 2 days after EOT (inclusive)
Recurrence rate | Up to 10 weeks
  Recurrence is defined as reappearance of diarrhea during the 8-week follow-up period.
Time to resolution of diarrhea | Up to 10 weeks
  Resolution of diarrhea (ROD) (≤ 3 unformed bowel movement (UBM) per day for at least 2 consecutive days) on study treatment and maintained for 2 days after end of treatment.

SECONDARY OUTCOMES:
Incidence of nephrotoxicity | Until 10 weeks
  Nephrotoxicity is defined as: serum creatinine increase of more than 0.5 mg/dL if the baseline serum creatinine was ≤ 3 mg/dL or a rise of > 1 mg/dL if the initial serum creatinine was > 3 mg/dL; or 50% increase from baseline; or a drop in calculated creatinine clearance using Cockroft-Gault formula of ≥ 50% from baseline.
Incidence of hepatotoxicit | Up to 10 weeks
  Hepatotoxicity is defined as: AST or ALT 3 times upper limit of normal or if AST or ALT baseline is abnormal, AST or ALT increase of ≥ 3 times the baseline and adverse events/ reactions using the MedDRA SMQ (Standardised MedDRA Query) "Hepatic Disorders".
Incidence of thrombocytopenia | Up to 10 weeks
  Thrombocytopenia is defined as: platelets < 100 000/mm3 or < 100 Giga/L
Incidence of hearing and balance/vestibular disorders | Up to 10 weeks
  Hearing and balance/vestibular disorders are defined as: identified via PT terms using MedDRA SMQ for "hearing and vestibular disorders" (narrow) and additionally the PT "balance disorder".
Additional renal endpoints: renal failure, dialysis and renal replacement therapy | Until 10 weeks
Any untoward adverse events/reactions | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- investigational site CHINA, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16229 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25280&tenant=MT_SNY_9011